CLINICAL TRIAL: NCT07066384
Title: Comparison of the Effectiveness of Breathing Yoga and Progressive Muscle Relaxation Techniques in Relieving Pain, Respiratory Complications and Kinesiophobia in Post-Liver Transplant Recipients
Brief Title: Comparison of Breathing Yoga and Progressive Muscle Relaxation Techniques After Transplantation
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Bitlis Eren University (Other)
Responsible Party: Principal Investigator, Serafettin Okutan, Principal Investigator, Assistant Professor Şerafettin OKUTAN, Surgical Nursing, Faculty of Health Sciences, Bitlis Eren University, Bitlis Eren University
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: okutan9
Record Dates: First submitted 2025-04-03; First posted 2025-07-15 (Actual); Last update posted 2025-09-18 (Actual); Status verified 2025-09

CONDITIONS: Breathing, Mouth; Muscle Relaxation; Pain, Postoperative; Kinesiophobia
Keywords: kinesiophobia; pain; breathing complications; breathing yoga; PMRTs
MeSH Terms: conditions — Mouth Breathing; Pain, Postoperative; Kinesiophobia; Pain

STUDY DESIGN:
Intervention Model Description: It will be conducted as a randomized controlled experimental study in a pretestpost- test control group experimental model.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- ıntervention group 1 (breathing yoga) (Experimental): Experimental group (Breathing Yoga):
  Data collection tools (patient introduction form, numerical rating scale, respiratory complications form, Tampa kinesiophobia scale) will be applied before the yoga breathing exercises intervention. Patients will be shown how to practice breathing yoga, and then they will be asked to do it. Breathing yoga consists of 6 stages.
  Patients will be given breathing yoga brochures. After discharge, patients will be asked to do breathing yoga once every 8 hours (3 times a day) for 3 months. Patients will be contacted by phone. For the application of the exercises, complications related to the disease, etc. After three months, patients will be invited to the outpatient clinic and during these outpatient clinic visits, scales and forms will be applied to these patients once again to collect posttest data.
  Interventions: Other: breathing yoga
- ıntervention group 2 (PMRTs) (Experimental): Experimental Group (Progressive Muscle Relaxation Techniques-PMRTs):
  Data collection tools (patient identification form, numerical rating scale, respiratory complications form, Tampa Kinesiophobia scale) will be applied before the progressive muscle relaxation exercise intervention. Progressive muscle relaxation exercises will be demonstrated to patients in practice, and then they will be asked to do them. PMRTs are applied to 11 different muscle groups.
  PMRTs brochures will be given to the patients. After the patients are discharged, they will be asked to perform PMRTs once every 8 hours (3 times a day) for 3 months. Patients will be contacted by phone. For the implementation of the exercises, complications related to the disease, etc. After three months, the patients will be invited to the outpatient clinic and during these outpatient clinic visits, the scales and forms will be applied to these patients once again to collect posttest data.
  Interventions: Other: PMRTs-Progressive Muscle Relaxation Techniques
- control group (No Intervention): Data collection tools (patient identification form, numerical rating scale, respiratory complications form, Tampa kinesiophobia scale) will be applied to the patients in the control group as part of the pretest. Patients with questions will be allowed to direct their questions to the researchers. After these questions are answered, no intervention will be made to the control group and the patients in the control group will not be contacted at any time for the next three months. After three months, the patients in the control group will be invited to the outpatient clinic and during these outpatient clinic visits, the scales and forms will be applied to these patients once again to collect posttest data.

INTERVENTIONS:
Other: breathing yoga — Yoga Breathing Exercises:
  1. Sama Vritti or "Equal Breathing":
  2. Abdominal Breathing Techniques:
  3. Nadi Shodhana or "Alternating Breathing":
  4. Kapalabhati or "Skull Shining Breath":
  5. Progressive Muscle Relaxation:
  6. Guided Visualization:
  Arms: ıntervention group 1 (breathing yoga)
Other: PMRTs-Progressive Muscle Relaxation Techniques — While patients are breathing in and out, tightening and releasing exercises are applied to 11 different muscle groups. It is applied for 15-20 minutes.
  Arms: ıntervention group 2 (PMRTs)

SUMMARY:
The study aims to compare the effectiveness of breathing yoga and progressive muscle relaxation techniques in relieving pain, respiratory complications and kinesiophobia in liver transplant recipients.

H1-0: Breathing yoga has no effect in reducing pain in liver transplant recipients.

H1-1: Breathing yoga has an effect in reducing pain in liver transplant recipients.

H2-0: Breathing yoga has no effect in reducing respiratory complications in liver transplant recipients.

H2-1: Breathing yoga has an effect in reducing respiratory complications in liver transplant recipients.

H3-0: Breathing yoga has no effect in relieving kinesiophobia in liver transplant recipients.

H3-1: Breathing yoga has an effect in relieving kinesiophobia in liver transplant recipients.

H4-0: PMRTs has no effect in reducing pain in liver transplant recipients.

H4-1: PMRTs have an effect on reducing pain in liver transplant recipients.

H5-0: PMRTs have no effect on reducing respiratory complications in liver transplant recipients.

H5-1: PMRTs have an effect on reducing respiratory complications in liver transplant recipients.

H6-0: PMRTs have no effect on relieving kinesiophobia in liver transplant recipients.

H6-1: PMRTs have an effect on relieving kinesiophobia in liver transplant recipients.

DETAILED DESCRIPTION:
Experimental group (Breathing Yoga):

Data collection tools (patient introduction form, numerical rating scale, respiratory complications form, Tampa kinesiophobia scale) will be applied before the yoga breathing exercises intervention. Patients will be shown how to practice breathing yoga, and then they will be asked to do it. The stages of breathing yoga are as follows:

Yoga Breathing Exercises:

1. Sama Vritti or "Equal Breathing":
2. Abdominal Breathing Techniques:
3. Nadi Shodhana or "Alternating Breathing":
4. Kapalabhati or "Skull Shining Breath":
5. Progressive Muscle Relaxation:
6. Guided Visualization:

Patients will be given breathing yoga brochures. After discharge, patients will be asked to do breathing yoga once every 8 hours (3 times a day) for 3 months. Patients will be contacted by phone. For the application of the exercises, complications related to the disease, etc. After three months, patients will be invited to the outpatient clinic and during these outpatient clinic visits, scales and forms will be applied to these patients once again to collect posttest data.

Experimental Group (Progressive Muscle Relaxation Techniques-PMRTs):

Data collection tools (patient identification form, numerical rating scale, respiratory complications form, Tampa Kinesiophobia scale) will be applied before the progressive muscle relaxation exercise intervention. Progressive muscle relaxation exercises will be demonstrated to patients in practice, and then they will be asked to do them. PMRTs stages are as follows:

The patient is placed in a semi-sitting/lying position in bed. While the patient is breathing in and out, 11 different muscle group tightening/releasing exercises are performed. PMRTs are performed by the researchers for 15-20 minutes on the patients. After PMRTs, patients are rested in a quiet and calm patient room.

PMRTs brochures will be given to the patients. After the patients are discharged, they will be asked to perform PMRTs once every 8 hours (3 times a day) for 3 months. Patients will be contacted by phone. For the implementation of the exercises, complications related to the disease, etc. After three months, the patients will be invited to the outpatient clinic and during these outpatient clinic visits, the scales and forms will be applied to these patients once again to collect posttest data.

Control group:

Data collection tools (patient identification form, numerical rating scale, respiratory complications form, Tampa kinesiophobia scale) will be applied to the patients in the control group as part of the pretest. Patients with questions will be allowed to direct their questions to the researchers. After these questions are answered, no intervention will be made to the control group and the patients in the control group will not be contacted at any time for the next three months. After three months, the patients in the control group will be invited to the outpatient clinic and during these outpatient clinic visits, the scales and forms will be applied to these patients once again to collect posttest data. After the data collection process is completed, breathing yoga and progressive muscle relaxation exercises will be demonstrated to the control group patients if they wish. It will be supported with brochures. Patients will be informed that they can contact the researchers by phone for information/support regarding the applications.

ELIGIBILITY:
Inclusion Criteria:

* Successful liver transplantation,
* Considered to be discharged after liver transplantation,
* Being 18 years old or older,
* No communication or language barriers,
* Agreeing to do PMRTs,
* Agreeing to do breathing yoga

Exclusion Criteria:

* Having any auditory or mental problems,
* Wanting to leave the study,
* Having difficulty/unable to do PMRTs,
* Having any joint-knee and orthopedic disorders,
* Having difficulty/unable to do breathing yoga.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 111 (Estimated)
Dates: Start 2025-03-01 (Actual); Primary Completion 2025-07-15 (Actual); Study Completion 2025-10-30 (Estimated)

PRIMARY OUTCOMES:
pain level | Discharged patients will be asked to perform breathing yoga/PMRT every 8 hours (three times a day) for three months. Posttest data will be collected at the end of the three months.
  Numerical Rating Scale (NRS):
  This scale, which is intended to determine the severity of pain, aims to have the patient describe their pain with numbers. In the form, 0 points are evaluated as "no pain", 1-3 points as "mild pain", 4-6 points as "moderate pain", and 7 and above points as "severe pain".

SECONDARY OUTCOMES:
Kinesiophobia level | Discharged patients will be asked to perform breathing yoga/PMRT every 8 hours (three times a day) for three months. Posttest data will be collected at the end of the three months.
  Tampa Kinesiophobia Scale (TKS):
  TKS is a 17-question questionnaire that has been validated and reliable in Turkish and is used to determine the presence of kinesiophobia. A 4-point Likert scoring system is used for each question in the scale. As a result of the survey, the person receives a total score between 17-68 according to the answers they give. A high score on the scale indicates that the person has high kinesiophobia.

CONTACTS AND LOCATIONS:
Overall Officials: Şerafettin OKUTAN, PhD., Principal Investigator — Bitlis Eren University
Locations (1):
- Bitlis Eren University, Bitlis, Turkey (Türkiye)